CLINICAL TRIAL: NCT06068426
Title: Incorporating Endoscopic Ultrasound and Elastography Towards Improving Outcomes of Pediatric Pancreatitis Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Vitale MD (Other)
Responsible Party: Sponsor-Investigator, David Vitale MD, Assistant Professor, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0499
Record Dates: First submitted 2023-06-26; First posted 2023-10-05 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pancreatitis; Acute Recurrent Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TUS SWE (Experimental): This arm includes two cohorts:
  1. Children with confirmed diagnosis of ARP or CP
  2. Controls (Children without a history of pancreatic disease)
  Interventions: Diagnostic Test: Transabdominal ultrasound Shear wave elastography

INTERVENTIONS:
Diagnostic Test: Transabdominal ultrasound Shear wave elastography — TUS SWE will be performed using a Canon Aplio i800 ultrasound system and a curved 1-6 MHz transducer. 2D SWE will be performed with measurement of shear wave speed in the head, body and tail of the pancreas.
  Other Names: TUS SWE

SUMMARY:
The main reason for this research study is to find out more about acute recurrent pancreatitis and chronic pancreatitis in children. There are few studies on childhood pancreatitis, so diagnosis and treatment are based on adult studies. This limits our understanding and treatment of these disorders in children.

Endoscopic ultrasound (EUS) is a tool used to assess and diagnose pancreatic disease. We can use ultrasound with shear wave elastography (SWE) to measure fibrosis (scarring) of the pancreas. We can use SWE on both EUS and transabdominal ultrasound (TUS) systems. Both TUS and EUS SWE have been studied for diagnosis of chronic pancreatitis in adult patients, however they have not been studied in children.

We plan to use EUS SWE and TUS SWE information in this study to help us understand pancreatitis in children. Children with pancreatitis and children without pancreatitis (controls) will be invited to participate in this study.

DETAILED DESCRIPTION:
The aims of the proposed study are as follows:

Aim 1: Characterize endoscopic ultrasound (EUS) findings of pediatric acute recurrent pancreatitis (ARP) and chronic pancreatitis (CP).

Adult criteria for EUS diagnosis of CP exist, but no such criteria exist for children. As such, the applicability of current diagnostic criteria to pediatric patients is unknown.

1.1: Catalogue grayscale EUS findings of ARP and CP in a pediatric cohort and compare to healthy controls. Hypothesis: EUS findings of ARP and CP in pediatric patients will differ from those of adult ARP and CP and will be characteristically different from healthy controls. Exp1: We will catalogue grayscale EUS findings in 40 pediatric

patients with known history of ARP or CP undergoing clinically indicated EUS and will compare those with findings in 20 patients without a history of pancreatitis who are undergoing EUS for other indications.

1.2: Benchmark grayscale EUS against other imaging modalities for diagnosis of CP, particularly early CP, in children. Hypothesis: Grayscale EUS findings will be more sensitive than other imaging modalities in all stages of CP. Exp2: We will test associations, in blinded fashion, of grayscale EUS findings catalogued under S.A1.1 in enrolled children with findings on alternative pancreas imaging modalities performed for clinical indications. Specifically, we will correlate to endoscopic retrograde cholangiopancreatography (ERCP), magnetic resonance cholangiopancreatography (MRCP) and computed tomography (CT) performed for clinical indications within +/- 3 months of the EUS.

Aim 2: Define the diagnostic performance of ultrasound elastography for CP and pancreatic stiffness as a measure of fibrosis in pediatric patients.

2.1: Define the diagnostic performance of EUS and TUS elastography for pediatric CP. Hypothesis: EUS and TUS elastography will have high specificity for CP with increased stiffness in patients compared to controls. Exp 1: Patients enrolled under Aim 1 will undergo shear wave elastography (SWE) measurement of the pancreas during EUS. These same patients will undergo research TUS with SWE of the pancreas. SWE results by both EUS and TUS will be evaluated for diagnostic performance for CP.

2.2: Define agreement between EUS and TUS measurement of pancreatic parenchymal stiffness in pediatric patients. Hypothesis: EUS and TUS measures of pancreatic parenchymal stiffness will agree with minimal bias. Exp2: EUS and TUS SWE data obtained under S.A2.1 will be evaluated for agreement and divergent cases will be investigated to define causes.

2.3: Define the diagnostic performance of elastography for pancreatic fibrosis. Hypothesis: SWE is a sensitive indicator of pancreatic fibrosis as identified by histology. Exp3: Patients undergoing clinically indicated total pancreatectomy and islet auto transplant (TPIAT) or other pancreatic surgical resection at our institution (approximately 20 per year) will be approached to undergo pre-operative TUS SWE. These SWE measurements, along with EUS SWE measurements obtained preoperatively, will be compared to binary and semi-quantitative assessments of pancreatic parenchymal fibrosis by histology.

ELIGIBILITY:
Pancreatitis Cohort:

Inclusion criteria:

* Confirmed diagnosis of ARP or CP by INSPPIRE criteria
* ≤ 21 years of age, male and female
* Children undergoing EUS for clinical care
* For Aim 2.3 only: Children undergoing TPIAT or other pancreatic resection

Exclusion criteria:

* Children <15 kg who cannot accommodate the size of endoscope
* Children with acute pancreatitis (AP) <6 weeks prior to EUS

Control Cohort:

Inclusion criteria:

* Children without a history of pancreatic disease undergoing EUS for other clinical indications
* ≤ 21 years of age, male and female

Exclusion criteria:

* Children <15 kg who cannot accommodate the size of endoscope
* Children with AP, ARP or CP

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Vitale, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Children With Confirmed Diagnosis of ARP or CP; Controls (Children Without a History of Pancreatic Disease): Transabdominal ultrasound Shear wave elastography: TUS SWE will be performed using a Canon Aplio i800 ultrasound system and a curved 1-6 MHz transducer. 2D SWE will be performed with measurement of shear wave speed in the head, body and tail of the pancreas.
Period: Overall Study
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Started | 45 | 21
Completed | 39 | 20
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Population: 45 subjects with ARP/CP were enrolled but only 39 completed the study. 21 controls were enrolled but only 20 completed the study. These 7 subjects were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease) | Total
Number analyzed (Participants) | 39 | 20 | 59
Age, Continuous [Mean (Full Range); unit: years] | 12.13 [6 to 19] | 15.1 [6 to 20] | 13.12 [6 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 20 | 11 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 32 | 19 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants] — Population: 7 subjects (6 with ARP/CP and 1 control) were enrolled but did not complete the study and were not evaluable. These 7 subjects were excluded from analysis.
  Participants
    United States | 39 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: EUS Pancreatic Findings- Rosemont Criteria
Description: Rosemont Criteria Features
  * Hyperechoic foci with shadowing (Major A)
  * Lobularity with honeycombing (Major B)
  * Lobularity without honeycombing (Minor)
  * Hyperechoic foci without shadowing (Minor)
  * Cysts (Minor)
  * Stranding (Minor)
  * Main pancreatic duct calculi (Major A)
  * Irregular main pancreatic duct contour (Minor)
  * Dilated side branches (Minor)
  * Main pancreatic duct dilation (Minor)
  * Hyperechoic main pancreatic duct margin (Minor)
Time Frame: At time of EUS procedure
Population: one test subject was excluded from the analysis because of unexpected findings of active acute pancreatitis at the time of the endoscopic ultrasound (EUS). This exclusion was necessary because acute pancreatitis can interfere with the evaluation of EUS findings related to chronic pancreatitis (CP) and acute recurrent pancreatitis (ARP).
Measure: Number; unit: percentage of participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 39 | 20
percentage of participants
  Hyperechoic foci with shadowing | 36 | 0
  Lobularity with honeycombing | 26 | 0
  lobularity without honeycombing | 36 | 20
  Hyperechoic foci without shadowing | 49 | 15
  Cysts | 10 | 0
  Stranding | 79 | 55
  Main pancreatic duct calculi | 10 | 0
  Irregular main pancreatic duct contour | 49 | 0
  Dilated side branches | 10 | 0
  Main pancreatic duct dilation | 15 | 0
  Hyperechoic main pancreatic duct margin | 36 | 0

2. Secondary Outcome: Calculated BMI
Description: Capturing weight(kg) and height(cm) to calculate
Time Frame: 6 months (3 months prior to endoscopic ultrasound through 3 months post-endoscopic ultrasound)
Population: BMI calculated from height and weight. Some participants did not have height and/or weight data available.
Measure: Median (Inter-Quartile Range); unit: kg/m2
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 38 | 15
kg/m2 | 21.3 [18.5 to 28.4] | 30.5 [23.7 to 35.9]

3. Secondary Outcome: Acute Recurrent Pancreatitis
Description: The presence or absence of recurrence of pancreatitis.
Time Frame: 6 months (3 months prior to endoscopic ultrasound through 3 months post-endoscopic ultrasound)
Population: This is a description of the number of subjects in the ARP/CP cohort who have been diagnosed with ARP. 0 Healthy controls would have ARP.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP
Number analyzed (Participants) | 39
Participants | 10

4. Secondary Outcome: Chronic Pancreatitis
Description: The presence or absence of Chronic pancreatitis diagnosis
Time Frame: 6 months (3 months prior to endoscopic ultrasound through 3 months post-endoscopic ultrasound)
Population: Description of the number of participants in the ARP/CP group with CP diagnosis. Healthy controls were not evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP
Number analyzed (Participants) | 39
Participants | 29

5. Secondary Outcome: Exocrine Pancreatic Insufficiency
Description: The presence or absence of exocrine pancreatic insufficiency diagnosis.
Time Frame: 6 months (3 months prior to endoscopic ultrasound through 3 months post-endoscopic ultrasound)
Population: A description of the presence or absence of exocrine pancreatic insufficiency diagnosis in the ARP/CP cohort. Healthy controls were also evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 39 | 20
Participants | 2 | 0

6. Secondary Outcome: Diabetes Mellitus
Description: The presence or absence of a diagnosis of diabetes.
Time Frame: 6 months (3 months prior to endoscopic ultrasound through 3 months post-endoscopic ultrasound)
Population: A description of the presence or absence of a diagnosis of diabetes in the ARP/CP cohort as well as healthy controls.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 39 | 20
Participants | 10 | 0

7. Secondary Outcome: EUS Rosemont Classification - Normal
Description: The Rosemont classification has been established to standardize an approach to EUS diagnosis of CP. The following criteria are used to determine the classification.
  Hyperechoic foci with shadowing Lobularity with honeycombing Lobularity without honeycombing Hyperechoic foci without shadowing Cysts Stranding Main pancreatic duct calculi Irregular main pancreatic duct contour Dilated side branches Main pancreatic duct dilation Hyperechoic main pancreatic duct margin
Time Frame: At time of EUS
Population: The number of subjects without any indications of CP based on Rosemont criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 39 | 20
Participants | 6 | 19

8. Secondary Outcome: EUS Rosemont Classification - Indeterminate for CP
Description: as for outcome 7
Time Frame: At time of EUS
Population: The number of participants with Indeterminate for CP based on Rosemont Criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 39 | 20
Participants | 11 | 1

9. Secondary Outcome: EUS Rosemont Classification - Suggestive of CP
Description: as for outcome 7
Time Frame: At time of EUS
Population: The number of participants with "Suggestive of CP" based on Rosemont Criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 39 | 20
Participants | 12 | 0

10. Secondary Outcome: EUS Rosemont Classification - Consistent With CP
Description: as for outcome 7
Time Frame: At time of EUS
Population: The number of participants with "Consistent with CP" based on Rosemont Criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 39 | 20
Participants | 10 | 0

11. Secondary Outcome: MRI Cambridge Grade: Normal
Description: Cambridge Grade:
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Severe)
Time Frame: At time of MRI
Population: The number of participants with "Normal" based on MRI Cambridge Grade criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 17 | 2
Participants | 4 | 2

12. Secondary Outcome: MRI Cambridge Grade: Equivocal
Description: Cambridge Grade:
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Severe)
Time Frame: At time of MRI
Population: The number of participants with "Equivocal" based on MRI Cambridge Grade criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 17 | 2
Participants | 0 | 0

13. Secondary Outcome: MRI Cambridge Grade: Mild
Description: Cambridge Grade:
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Severe)
Time Frame: At time of MRI
Population: The number of participants with "Mild" based on MRI Cambridge Grade criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 17 | 2
Participants | 0 | 0

14. Secondary Outcome: MRI Cambridge Grade: Moderate
Description: Cambridge Grade:
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Severe)
Time Frame: At time of MRI
Population: The number of participants with "Moderate" based on MRI Cambridge Grade criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 17 | 1
Participants | 5 | 0

15. Secondary Outcome: MRI Cambridge Grade: Severe
Description: Cambridge Grade:
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Marked)
Time Frame: At time of MRI
Population: The number of participants with "Severe" based on MRI Cambridge Grade criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
Number analyzed (Participants) | 17 | 2
Participants | 8 | 0

16. Secondary Outcome: ERCP Cambridge Criteria: Normal
Description: Cambridge Criteria
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Marked)
Time Frame: At time of ERCP
Population: The number of participants with "Normal" based on ERCP Cambridge Criteria. Healthy controls were not analyzed here.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP
Number analyzed (Participants) | 28
Participants | 0

17. Secondary Outcome: ERCP Cambridge Criteria: Equivocal
Description: Cambridge Criteria
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Marked)
Time Frame: At time of ERCP
Population: The number of participants with "Equivocal" based on ERCP Cambridge Criteria. Healthy controls were not analyzed here.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP
Number analyzed (Participants) | 28
Participants | 4

18. Secondary Outcome: ERCP Cambridge Criteria: Mild
Description: Cambridge Criteria
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Marked)
Time Frame: At time of ERCP
Population: The number of participants with "Mild" based on ERCP Cambridge Criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP
Number analyzed (Participants) | 28
Participants | 1

19. Secondary Outcome: ERCP Cambridge Criteria: Moderate
Description: Cambridge Criteria
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Marked)
Time Frame: At time of ERCP
Population: The number of participants with "Moderate" based on ERCP Cambridge Criteria. Healthy controls were not analyzed here.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP
Number analyzed (Participants) | 28
Participants | 8

20. Secondary Outcome: ERCP Cambridge Criteria: Marked
Description: Cambridge Criteria
  1. (Normal)
  2. (Equivocal)
  3. (Mild)
  4. (Moderate)
  5. (Marked)
Time Frame: At time of ERCP
Population: The number of participants with "Marked" based on ERCP Cambridge Criteria. Healthy controls were not analyzed here.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Confirmed Diagnosis of ARP or CP
Number analyzed (Participants) | 28
Participants | 15

ADVERSE EVENTS:
Time Frame: At time of EUS procedure and at time of MRCP or CT imaging
Description: Per the IRB approved study protocol: "Adverse events related to the study procedures will be monitored by the study coordinator and reported to the PI. The PI will then report any adverse events in writing to the CCHMC IRB within the time frame specified in the IRB guidelines."
  Only adverse events related to study procedures would be reported. No adverse events were reported.
Arm/Group | Children With Confirmed Diagnosis of ARP or CP | Controls (Children Without a History of Pancreatic Disease)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/21
Other Adverse Events (participants affected / at risk) | 0/45 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT06068426/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT06068426/ICF_001.pdf